CLINICAL TRIAL: NCT03340246
Title: Delayed or Immediate Local Treatment of Varicose Veins
Brief Title: Delayed or Immediate Local Treatment of Veins
Acronym: DELICATVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maarit Venermo, Professor of Vascular Surgery, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DELICATVE
Record Dates: First submitted 2017-10-13; First posted 2017-11-13 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Varicose Veins Leg
Keywords: Varicose veins, phlebectomy
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate phlebectomy (Active Comparator): Mechanochemical ablation of main trunk and immediate phlebectomy of varicosities
  Interventions: Procedure: Immediate phlebectomy
- Delayed treatment (Experimental): Mechanochemical ablation of main trunk. Evaluation of varicosities at 3 months with sclerotherapy if required
  Interventions: Procedure: Delayed sclerotherapy

INTERVENTIONS:
Procedure: Delayed sclerotherapy — See arm descriptions
  Arms: Delayed treatment
Procedure: Immediate phlebectomy — See arm description
  Arms: Immediate phlebectomy

SUMMARY:
Varicose veins affect a majority of adult patients and cause a decreased quality of life. In recent years, standard practice has been to perform thermoablation and local phlebectomies in the same procedure. There is conflicting data on the long-term outcome of the local varicose veins; there seems to be a need for more re-interventions if the local varicosities are not treated immediately. On the other hand, the prolonged combined procedure increases procedural pain and bleeding, as well as the risk for complications from deep vein thrombosis/pulmonary embolism.

This trial aims to evaluate the need for immediate treatment of local varicosities and the potential sufficiency of main trunk treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound verified insufficiency of great saphenous vein (GSV)
* GSV diameter 5-10 mm
* C2-C4 varicosities
* Most proximal insufficient branch in the distal thigh
* Written and signed informed consent

Exclusion Criteria:

* Peripheral arterial disease
* Body mass index >40
* Lymphoedema
* Known allergy to sclerosant
* Any known coagulopathy or history of deep vein thrombosis
* Severe illness
* Pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-05-04 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Need for sclerotherapy | 3 months
  Need for sclerotherapy of varicosities at three months after ablation of main trunk. Evaluated by the CEAP-classification of venous insufficiency. >C2 will be eligible for treatment.

SECONDARY OUTCOMES:
Patient satisfaction | 3 months
  Overall patient satisfaction and symptoms regarding varicosities and procedure at three months. Evaluated by the Aberdeen Varicose Veins Questionnaire (AVVQ). The AVVQ is a validated test, in which patients are asked to check boxes with regard to symptoms and quality of life (QoL). Scale 0-100, with 100 indicating worst possible QoL.
Occlusion rate of great saphenous vein | 36 months
  Long-term occlusion rate of main trunk after mechanochemical ablation, evaluated by duplex ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Karoliina Halmesmäki, M.D., Ph.D, Principal Investigator — Helsinki University Central Hospital; Maarit Venermo, M.D., Ph.D., Study Director — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided